CLINICAL TRIAL: NCT05683028
Title: Cognitive Remediation Following Electroconvulsive Therapy in Patients with Treatment Resistant Depression: Randomized Controlled Trail of an Intervention for Relapse Prevention
Brief Title: RCT for Electroconvulsive Treatment Followed by Cognitive Control Training
Acronym: ECT-CCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); King Baudouin Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-1089
Record Dates: First submitted 2020-03-16; First posted 2023-01-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depressive Episode; Electroconvulsive Therapy; Cognitive Remediation
Keywords: Cognitive control training

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either intervention or placebo.
Who Masked: Participant, Outcomes Assessor
Masking Description: Upon registration in the computer-based training, the computer will randomly allocate participants to either cognitive control training or placebo condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive control training (Experimental): Cognitive Control Training (CCT) makes use of a very basic cognitive task that strongly loads on working memory and cognitive control processes, namely the adaptive Paced Auditory Serial Addition Task (aPASAT) where participants are given a number every 3 seconds and are asked to add the number they just heard with the number they heard before. Task difficulty is modified based on the participants current task performance, allowing training of cognitive control. Participants in the intervention group will start the CCT training after completion of ECT with a maximum time interval of 7 days. Training sessions will be performed on a tablet or computer and participants will complete five sessions per week (20 minutes per session) for a period of two weeks.
  Interventions: Behavioral: Cognitive Control Training
- Active Control (Active Comparator): Participants in the active control group will start placebo training after completion of ECT with a maximum time interval of 7 days. The placebo task consists of a task similar to the experimental condition but that does not train cognitive control. Prior research confirmed that this condition controls for non-specific effects of the training and motivational issues. Participants will perform the sessions on a tablet or computer and complete five sessions per week (20 minutes per session) for a period of two weeks.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Cognitive Control Training — Cognitive Control Training (CCT) makes use of a very basic cognitive task that strongly loads on working memory and cognitive control processes, namely the adaptive Paced Auditory Serial Addition Task (aPASAT) where participants are given a number every 3 seconds and are asked to add the number they just heard with the number they heard before. Task difficulty is modified based on the participants current task performance, allowing training of cognitive control. Participants in the intervention group will start the CCT training after completion of ECT with a maximum time interval of 7 days. Training sessions will be performed on a tablet or computer and participants will complete five sessions per week (20 minutes per session) for a period of two weeks.
  Other Names: aPASAT
  Arms: Cognitive control training
Behavioral: Active Control — Participants in the active control group will start placebo training after completion of ECT with a maximum time interval of 7 days. The placebo task consists of a task similar to the experimental condition but that does not train cognitive control. Prior research confirmed that this condition controls for non-specific effects of the training and motivational issues. Participants will perform the sessions on a tablet or computer and complete five sessions per week (20 minutes per session) for a period of two weeks.
  Arms: Active Control

SUMMARY:
Major depressive disorder (MDD) is worldwide one of the most prevalent and disabling mental health conditions. Electroconvulsive therapy (ECT) is a safe and effective treatment even though 6-month relapse rates are high. Cognitive side effects of ECT, such as reduced cognitive control, might trigger mechanisms that increase relapse in patients. As such, cognitive control training (CCT) holds promise as a non-pharmacological strategy to improve long-term effects of ECT (i.e., increase remission, and reduce depression relapse).

DETAILED DESCRIPTION:
Eighty-eight participants aged between 18-70 years with major depressive disorder who start electroconvulsive treatment (ECT) will be included in this randomized controlled trial (RCT). Following (partial) response to ECT treatment (at least a 25% reduction of clinical symptoms), participants will be randomly assigned to a computer based CCT or active placebo control. A first aim of this RCT is to assess the effects of CCT compared to an active placebo condition on depression symptomatology, cognitive complaints, and quality of life. Secondly, participants will be monitored every two weeks for a period of six months following CCT/active placebo, allowing the detection of potential relapse of depression. Thirdly, the investigators will assess participant evaluation of the addition of cognitive remediation to ECT using qualitative interview methods (satisfaction, acceptability and appropriateness). Finally, in order to further advance our understanding of the mechanisms underlying effects of CCT, exploratory analyses may be conducted using facial video footage collected during the CCT/active control phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 70 years old
* current major depressive episode with treatment resistance
* eligibility and consent for ECT treatment
* ability to provide consent to study

Exclusion Criteria:

* neurodegenerative disorder or MOCA < 18
* catatonia
* schizophrenia
* alcohol use disorder in previous year
* prior ECT treatment
* insufficient computer knowledge or analphabetism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Change in severity of depressive symptoms, clinician-rated (HAM-D) | 1-7 days before first ECT session, 1-7 days post ECT completion, 1-7 days after intervention/placebo completion, 3 months after ECT completion, and 6 months after ECT completion
  The Hamilton Depression Rating Scale (HAM-D) is a clinician rated questionnaire with 17 items scored on a three or five-point Likert-type scale. Amongst other symptoms of depression, items include mood, insomnia and suicidal ideations. Higher scores indicate increased severity of depression with a maximum score of 50 and minimum of 0.
Change in severity of depressive symptoms, self-reported (BDI-II) | 1-7 days before first ECT session, 1-7 days post ECT completion, 1-7 days after intervention/placebo completion, 3 months after ECT completion, and 6 months after ECT completion
  The Beck Depression Inventory (BDI-II) is a 21-item self-report questionnaire regarding symptoms of depression with good validity and reliability. Higher scores indicate increased severity of depression. Minimum score is 0 and 63 is the maximum score.
Change in depressive symptoms and quality of life, self-reported (RDQ) | 1-7 days before first ECT session, 1-7 days post ECT completion, 1-7 days after intervention/placebo completion, 3 months after ECT completion, and 6 months after ECT completion
  The Remission from Depression Questionnaire (RDQ) will inform about seven domains: symptoms of depression, non-depressive symptoms, features of positive mental health, coping ability, functioning, life satisfaction and a general sense of well-being. The RDQ is a 41-item questionnaire. Higher scores indicate increased severity of depression. Minimum score is 0 and 82 is the maximum score.

SECONDARY OUTCOMES:
Subjective memory complaints (SSMQ) | 1-7 days before first ECT session, 1-7 days post ECT completion, 1-7 days after intervention/placebo completion, 3 months after ECT completion, and 6 months after ECT completion
  To assess subjective cognitive functioning the Dutch version of the Squire Subjective Memory Questionnaire (SSMQ) (Squire, Wetzel et al. 1979) will be administered. this is a self-report questionnaire consisting of 18 items. The patients' answers are scored between -4 (worse than before), 0 (same as before), and +4 (better than before) points, the sum of which are added together to obtain a final score. A negative score shows an increase in the degree of forgetfulness.
Quality of Life in Depression Scale (QLDS) | 1-7 days before first ECT session, 1-7 days post ECT completion, 1-7 days after intervention/placebo completion, 3 months after ECT completion, and 6 months after ECT completion
  This 34-item questionnaire, developed by qualitative interviews, asks patients to rate statements regarding fulfillment of universal human needs such as 'I take good care of myself' and 'I like to know what is going on in the world'.
Rumination (RRS-10) | 1-7 days before first ECT session, 1-7 days post ECT completion, 1-7 days after intervention/placebo completion, 3 months after ECT completion, and 6 months after ECT completion
  The Ruminative Response Scale (RRS-10) will be used to monitor rumination or repetitive negative thinking as this is a well-established cognitive risk factor for MDE. This patient-rated scale consists of 10 items. A higher score indicates a higher degree of rumination with a minimum score of 10 and maximum score of 40.
Cognition (CANTAB) | 1-7 days before first ECT session, 1-7 days post ECT completion, 1-7 days after intervention/placebo completion, 3 months after ECT completion, and 6 months after ECT completion
  Pattern Recognition Memory (measuring visual pattern recognition memory) and One Touch Stockings of Cambridge (measuring spatial spanning and working memory). A third test, Motor Screening was included to measure general sensorimotor skills.
Cognition (Paced Auditory Serial Addition Task - PASAT) | 1-7 days before first ECT session, 1-7 days post ECT completion, 1-7 days after intervention/placebo completion, 3 months after ECT completion and 6 months after ECT completion
  Neuropsychological test to assess capacity and rate of information processing as well as sustained and divided attention.
Acceptability and satisfaction | 1 - 30 days after CCT training completion
  Qualitative interviews will be conducted with a maximum of 20 patients and family members to explore acceptability of the ECT procedure and the intervention.
Time to relapse | Up to 6 months monitoring
  By decreasing depression symptomatology we expect a decrease in relapse rates and a prolonged time-to-relapse-interval as measured by telephone interviews, once every two weeks, in patients who achieve remission.
Facial features from video footage | 2 weeks during CCT or placebo intervention
  During CCT or placebo training facial video footage will be collected from which different facial features will be extracted with the use of automated algorithms. These facial features could give insight into working processes during cognitive training versus placebo training. Certain facial features have shown to be indicative of learning, engagement and depressive symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Lemmens, MD, PhD, Study Director — UZGhent; Marie-Anne Vanderhasselt, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available due to confidentiality issues but are available from the corresponding author upon reasonable request.